CLINICAL TRIAL: NCT02288728
Title: Remnant Stomach-jejunum Double Tract Anastomosis vs. Gastric Tube Anastomosis to Proximal Gastrectomy of Early Gastric Cancer- a Randomized Controlled Trial
Brief Title: Double Tract Anastomosis and Gastric Tube Anastomosis to Proximal Gastrectomy
Acronym: DTA&GTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough paticipants enroll in this study.
Sponsor: Jian-Kun Hu (Other)
Responsible Party: Sponsor-Investigator, Jian-Kun Hu, Vice director of the Gastrointestinal Surgery Derpartment, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH-GC-01
Record Dates: First submitted 2014-09-29; First posted 2014-11-11 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Complications; Quality of Life; Remnant Gastritis; Reflux Esophagitis
Keywords: Proximal gastrectomy; quality of life; mortality; morbidity
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (double-track anastomosis) (Experimental): Patients in the Group B will received the double-track anastomosis with proximal gastrectomy.
  Interventions: Procedure: Double-track anastomosis
- Group A (Gastric tube anastomosis) (Other): Patients in the Group A (Gastric tube anastomosis) will take the gastric tube anastomosis with proximal gastrectomy.
  Interventions: Procedure: Gastric tube anastomosis

INTERVENTIONS:
Procedure: Gastric tube anastomosis — In the gastric tube group, the lesser curvature of the gastric remnant approximately 3 cm proximal to the pylorus was removed first by a linear stapling device. An approximately 5-cm-wide tubular stomach was then constructed with preserved right gastric vessels. The length of the tube was consistent with the greater curvature of the residual stomach. The reconstructed gastric tube was lastly anastomosed with the proximal esophageal end.
  (Reference: Chen XF, Zhang B, Chen ZX, Hu JK, Dai B, Wang F, Yang HX, Chen JP. Gastric tube reconstruction reduces postoperative gastroesophageal reflux in adenocarcinoma of esophagogastric junction. Dig Dis Sci. 2012;57(3):738-745.)
  Arms: Group A (Gastric tube anastomosis)
Procedure: Double-track anastomosis — Double-track anastomosis group: First, cut off the jejunum about 15-20 cm away from the Treitz ligament; Second, Roux-en-Y esophagojejunostomy (E-J stomy, first anastomosis) was perform by 25mm circular stapler device; Third, from 30-40cm to the E-J stomy, perform the side-to-side gastrojejunostomy (G-J stomy, second anastomosis). Forth, from 25-30cm to the G-J stomy, perform the jejunojejunostomy (J-J stomy, third anastomosis).
  (Reference: Ahn SH, Jung do H, Son SY, Lee CM, Park do J, Kim HH. Laparoscopic double-tract proximal gastrectomy for proximal early gastric cancer. Gastric Cancer. 2014;17(3):562-70.)
  Arms: Group B (double-track anastomosis)

SUMMARY:
Gastric cancer as one of the most common gastrointestinal cancers, radical resection of primary lesions combined with dissection of regional lymph-nodes is acknowledged by surgeons all over the world. When compared with the advanced upper third gastric cancer, proximal gastrectomy has been acknowledged as the standard therapeutic strategy for the early gastric cancer located in the upper third of the stomach. However, due to abandon the anti-reflux barrier of the digestive system caused by the dissection of the cardia and the lower esophageal sphincter, the belching、hiccup、Acid reflux、heartburn、chest pain symptoms and as well as the reflux esophagitis caused by the traditional esophagostomy permanently influence the postoperative quality of life for those patients. Nowadays, relationship between the digestive track reconstruction for proximal gastrectomy and the postoperative quality of life is still with controversies. Previous study reported the gastric tube anastomosis can minimize the reflux related symptoms when compared with traditional esophagogastrostomy. There still exited some patients need long-term anti-acid drug to control the reflux symptoms although underwent the gastric tube anastomosis. The double-track anastomosis for proximal gastrectomy may successfully control the reflux symptoms and there existed study found it is as safe as the esophagostomy. But there has no randomized control study to compare the postoperative quality of life between the gastric tube anastomosis and double-track anastomosis for proximal gastrectomy.

By the reasons above, a randomized controlled trial is conducted with the intention to compare the intraoperative and postoperative mortality and morbidity and the postoperative quality of life between the esophagogastrostomy and the double-track anastomosis in the proximal gastrectomy for gastric cancer patients.

DETAILED DESCRIPTION:
Standard Operating Procedure (SOP)

1. Preoperative evaluation Patients satisfied with inclusion/exclusion criteria will be informed to join in the clinical study and signature the inform consent.
2. Randomization: Intraoperative evaluation found that R0, proximal gastrectomy can be performed, the case will entrance into the Randomization period. Random numbers are computer-generated, with the third party applications.
3. Surgical procedures: The surgical treatments is adopted the proximal gastrectomy according to the Japanese Gastric Cancer treatments guidelines, 2010, Version 3. Group A take the gastric tube anastomosis and Group B take the double-track anastomosis (the reconstruction method is described in the intervention section of study groups). The two study will take the similar surgical procedures except for the digestive track reconstruction.
4. Postoperative recovery: Postoperative recovery period need to collect those relevant parameters of all the patients. All the relevant parameters had definitely definition in the Case Report Form of this study which included the preoperative, intraoperative and postoperative clinicopathologic characteristics.
5. Follow-up: The follow-up of this study divide into two parts, the postoperative quality of life and tumor characteristics outcomes. The information of the postoperative quality of life is collected by the European Organization for Research and Treatment of Cancer (EORCT) QLQ-C30 and STO-22 questionnaires. At the postoperative 12 moths, the upper gastrointestinal scope is needed to examine the reflux esophagitis and the remnant gastritis according to Los Angeles Classification of esophagitis. The tumor related outcomes included long-term postoperative complications, recurrence type, relapse free survival (months) and the overall survival (months).

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed upper third gastric adenocarcinoma, and predictively feasible of proximal gastrectomy ;
2. Predictively resectable diseases, early gastric cancer, of preoperative staging JGCA 14th Edition cT1N0M0-T2N0M0;
3. Age：≤75 years, or ≥18 years;
4. Without serious disease and malignance disease;
5. Patients without previous history of upper abdominal surgery;
6. WHO performance score ≤2, ASA score ≤3;
7. No limit to sexual and race;
8. informed consent required.

Exclusion Criteria:

1. With the history of the malignance disease;
2. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc.
3. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
4. Severity mental diseases;
5. After signature the Clinical trial agreement, patients and their agent will quit the trial;
6. primary lesion cannot be resected in the pattern of transabdominal proximal gastrectomy, but for total gastrectomy, Whipple's procedure, or combined organ resection or with a transthoracic approach surgery
7. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
postoperative mortality and morbidity | postoperative period (30 days)

SECONDARY OUTCOMES:
Intraoperative mortality and morbidity | Intraoperative
postoperative quality of life | Postoperative period (at least one year)
remnant gastritis | postoperative period (one year)
  Evaluated by Los Angeles classification. Reference: Lundell LR, Dent J, Bennett JR, et al. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut 1999; 45: 172-80.
reflux esophagitis | Postoperative period (one year)
  Evaluated by Los Angeles classification. Reference: Lundell LR, Dent J, Bennett JR, et al. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut 1999; 45: 172-80.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China